CLINICAL TRIAL: NCT04366453
Title: Evaluation of the Ejection Fraction of the Left Ventricle in the Emergency Room by a New Automatic Evaluation Tool in a Pocket Ultrasound Scanner: A Reproducibility Study
Brief Title: Evaluation of LVEF by a New Automatic Evaluation Tool in a Pocket Ultrasound Scanner
Acronym: ReproAuto_FEVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2019/XB-01; 2019-A03140-57 (Other: RCB number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Echocardiography; Medicine, Emergency; Technology Assessment, Biomedical; Heart Diseases
MeSH Terms: conditions — Emergencies; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echocardiography (Other): • Echocardiography performed by the evaluator 1: 2 LVEF visual evaluations 2 LVEF automatic evaluations
  • Echocardiography performed by the evaluator 2: 2 LVEF visual evaluations 2 LVEF automatic evaluations
  Interventions: Procedure: echocardiography

INTERVENTIONS:
Procedure: echocardiography — Four measurements in echocardiography performed in addition to standard care

SUMMARY:
Clinical ultrasound has become essential in emergency medicine. The guidelines are to use of echocardiography in specific contexts: dyspnea, hypotension or chest pain. The evaluation of left ventricle ejection fraction (LVEF) is one of the basic objectives of echocardiography. The reference assessment in emergency medicine is visual assessment. It suffers from poor inter-observer reproducibility. Pocket ultrasound scanners seem to meet the constraints of point-of-care ultrasound. A new tool is available on a pocket ultrasound device: the automatic evaluation of LVEF. Its interest could be to have a better inter-observer reproducibility than visual evaluation.

ELIGIBILITY:
Inclusion criteria:

* Patient over 18 years of age
* Management in the investigator centre
* Admitted for dyspnea or hypotension or chest pain

Exclusion criteria:

* Age < 18 years
* Patient not benefiting from a social security system
* Patient deprived of liberty
* Patient under the protection of justice, under guardianship or curatorship
* Patient refusing to participate in the study
* Inability to provide the patient with informed information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
evaluate the interobserver reproducibility | Day 0
  evaluate the interobserver reproducibility of the automatic measurement of LVEF with a pocket ultrasound device

SECONDARY OUTCOMES:
Assess the interobserver reproducibility of visual LVEF | day 0
  Assess the interobserver reproducibility of visual LVEF
Interobserver reproducibility of the visual LVEF measurement; | Day 0
  Assess the interobserver reproducibility of the visual LVEF measurement;
Evaluate the intraobserver reproducibility of the automatic LVEF measurement | Day 0
  Evaluate the intraobserver reproducibility of the automatic LVEF measurement
Ability of the pocket ultrasound scanner to give an ultrasound image useable by the doctor performing the examination. | Day 0
  Compare the feasibility of each method (visual and automatic) to obtain an ultrasound image useable by the doctor performing the examination.
Ability of the pocket ultrasound scanner to give an ultrasound image useable by the doctor performing the examination considering image quality | Day 0
  Evaluation of Image quality obtained by each méthod (Visual and Automatic)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bobbia, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No